CLINICAL TRIAL: NCT02185690
Title: A Phase I/Ib Study of MEK162, a MEK Inhibitor, in Combination With Carboplatin and Pemetrexed in Patients With Non-squamous Carcinoma of the Lung
Acronym: MEK162
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162ACA02T; CMEK162ACA02T (Other: Novartis Pharmaceuticals Canada Inc)
Record Dates: First submitted 2014-04-09; First posted 2014-07-09 (Estimated); Results first posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Lungcancer
Keywords: Lung cancer; Non small cell lung cancer; non squamous; pemetrexed; carboplatin; binimetinib; chemotherapy; combination chemotherapy; Phase 1; Princess Margaret Cancer Centre; carcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — binimetinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Binimetinib efficacy/safety (Other): This is a Phase I/Ib, open-label, dose-escalation, multi-center, non-randomized study designed to evaluate the safety and tolerability of oral Binimetinib in combination with carboplatin and pemetrexed.
  Phase I part A standard 3+3 dose-escalation will be used to determine the maximum administered dose (MAD) and the RP2D for the combination in subjects with advanced non-squamous lung carcinoma.
  Phase Ib part Once RP2D has been identified, an expansion cohort will be accrued; these patients will be stratified by KRAS genotype.
  The RP2D will be expanded by enrolling additional patients, stratified by KRAS genotype, to a total of 30 patients eligible for the safety set (including those treated at the same dose combination in the dose-escalation phase of the study who are eligible for the safety set) to be evaluated for safety, tolerability, pharmacokinetics and biologic activity of MEK162.
  Interventions: Drug: Binimetinib; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Binimetinib — Continuous MEK162 with dose escalation until the Recommended Phase 2 dose (RP2D) one dose level below the Maximum administered dose (MAD) or progression of disease.
  MEK162 tablets 15 mg strength will be taken orally on a BID dose schedule.
  Other Names: MEK162
Drug: Pemetrexed — 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Other Names: Alimta
Drug: Carboplatin — 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Other Names: Paraplatin AG

SUMMARY:
MEK162 has shown significant inhibition of tumor growth as a single agent in NSCLC xenograft models in mice and human cancer cells in vitro, which have KRAS and/or other mutations. These data suggest that MEK162 may provide a potential benefit in cancer indications harboring these mutations. MEK162 is currently being investigated in phase I clinical testing and has been well tolerated up to an MTD of 45mg BID in cancer patients.

There has been little change in survival benefit for patients with non-small cell lung cancer in recent years. Emerging new treatment options relying on molecular and genetic markers are being studied extensively. Thus, there has been a shift to manage non-small cell lung cancer with molecular targeted therapies in combination with standard chemotherapy. This study will be targeting patients with KRAS mutations.

DETAILED DESCRIPTION:
OBJECTIVES

1.1 Primary Objectives

* To assess the safety of MEK162 administered in combination with carboplatin and pemetrexed as first line treatment in advanced non-small cell lung cancer (NSCLC).
* To determine the recommended phase II dose (RP2D) of MEK162 to be used when given in a continuous dosing schedule together with pemetrexed and carboplatin administered on a 3-weekly schedule as first line treatment in advanced NSCLC.
* To explore the efficacy (as measured by tumor response in the Phase Ib portion) of the combination of MEK162 in addition to pemetrexed and carboplatin in treatment-naïve patients with EGFR wild-type, ALK-rearrangement negative NSCLC of the lung.

1.2 Secondary Objectives

* To characterize the population pharmacokinetics of MEK162 administered in combination with carboplatin and pemetrexed (Phase I).
* To explore relationships between KRAS mutation (and sub-types) and additional genomic mutations and objective clinical response.

1.3 Trial End-points Primary Phase I • Development of dose-limiting toxicity (DLT), (defined in section 4.3) as measured with NCI CTC AE v4.

Phase Ib

• Objective response rate (ORR) as per RECIST v1.1.

Secondary Phase I • Adverse events, serious adverse events, changes in hematology and chemistry values, vital signs, ECGs.

Phase Ib

* Evaluation of response rate (RR), progression-free survival (PFS) and disease control rate (DCR) for patients with and without KRAS mutation in tumor tissue.
* Exploratory analysis of KRAS mutation sub-type.

Exploratory end-points

• A limited sampling strategy pharmacokinetic model will be used to ensure that the clearance of MEK162 is not influenced by the concurrent administration of pemetrexed-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for enrolment on the study must meet all of the following criteria:
* Patients with histologically confirmed non-squamous EGFR wild-type, ALK-rearrangement negative carcinoma of lung. Patients with neuroendocrine carcinoma, mixed small and non-small cell carcinoma or squamous carcinoma are not eligible.
* Tissue available for KRAS mutation status analysis.
* Patients must have metastatic disease (Incurable stage IIIB/stage IV).
* Patients must have clinically and/or radiographically documented measurable disease. At least one site of disease must be unidimensionally measurable by RECIST v1.1 as follows (Eisenhauer et al.):

CT-scan, physical exam ≥10 mm Chest X-ray ≥20 mm Lymph node short axis ≥15 mm

* All radiology studies must be performed within 28 days prior to registration (35 days if negative).
* Lesions in previously irradiated areas should not be selected unless there is clear evidence of progression in such lesions.
* Patients may not have received any prior systemic treatment for metastatic NSCLC. Patients who have received adjuvant treatment or chemoradiation for stage III disease should have completed this ≥12 months prior to study enrollment.
* Patients with stable CNS metastases are permitted if stability of disease is documented with imaging ≥28 days after treatment completion, are and off corticosteroids by day 1 of study treatment.
* Patients may have had prior malignancy if definitively treated and/or, in the opinion of the investigator, the only active malignancy is NSCLC. Patients with mixed small cell lung cancer histology are excluded. Patients who have received radiotherapy to >30% bone marrow are excluded. Consult PI if unsure whether second malignancies meet requirements specified above.
* In patients treated for other malignancy, all prior treatment-related toxicities must be CTCAE v4.0 ≤ Grade 1 (except alopecia) at the time of enrollment.
* Able to swallow and retain oral medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Patients receiving medications or substances that are inhibitors or inducers of CYP1A2, CYP2A19, CYP2B6, CYP3A4 and/or UGT1A1 and UGT1A9 are eligible but these drugs must be used with caution (Appendix C).

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx;

* Patients must be aged ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ and laboratory parameters, defined below.
* Laboratory Requirements - within 7 days prior to enrollment:

Haematology: absolute granulocytes ≥1.5 × 109/L platelets ≥100 × 109/L Biochemistry: bilirubin ≤1.25 × institutional upper limit of normal AST(SGOT) ≤2.5 × institutional upper limit of normal /ALT(SGPT) or ≤5 × institutional upper limit of normal in the presence of liver metastases

creatinine clearance ≥45 mL/min/1.73 m2

-Patients must be able to provide Informed Consent based on the details below:

* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR):

  * History of RVO or CSR, or predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled systemic disease such as hypertension, diabetes mellitus, or history of hyperviscosity or hypercoagulability syndromes). Patients with prior deep venous thrombosis or pulmonary embolism are permitted.
  * Visible retinal pathology as assessed by ophthalmologic exam that is considered a risk factor for RVO or CSR such as:
* Evidence of new optic disc cupping
* Evidence of new visual field defects on automated perimetry
* Intraocular pressure >21mmHg as measured by tonography
* Any serious and/or unstable pre-existing medical (aside from malignancy exception), psychiatric disorder, or other conditions that could interfere with subjects' safety, obtaining informed consent or compliance to the study procedures, in the opinion of the PI.
* History of interstitial lung disease or pneumonitis.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal metabolic or cardiac disease).
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events (e.g. congenital long QT syndrome, family history of long QT syndrome, hypokalemia) or baseline QTcB interval ≥480 msec.
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within the past 6 months or cardiac metastases.
* History or evidence of current clinically significant uncontrolled arrhythmias.
* History or evidence of current ≥Class II congestive heart failure as defined by New York Heart Association (NYHA).
* Known positivity for Hepatitis B surface antigen or Hepatitis C antibody.
* Known Human Immunodeficiency Virus (HIV) infection.
* Treatment refractory hypertension defined as a blood pressure systolic >140 mmHg and/or diastolic >90 mmHg which cannot be controlled by anti-hypertensive therapy.
* Subjects with intra-cardiac defibrillators or permanent pacemakers.
* Pregnant or nursing (lactating) women are excluded.
* Female patient of child bearing potential must have a negative serum or urine pregnancy test.
* Women of child-bearing potential must agree to use of appropriate contraceptive methods throughout the study and for 120 days after, These methods include
* Total abstinence or 2 barrier methods or a barrier method plus hormonal method from visit 1 to 120 days after the last dose of treatment.
* Men must agree to use an appropriate method of contraception starting with first dose of study drug through 120 days after the last dose of treatment (see above).
* Whilst not excluded, patients with significant impaired hearing must be made aware of potential ototoxicity and may choose not to be included. If included, baseline audiograms are recommended and should be followed by repeat audiograms prior to cycle 2.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, MD, Principal Investigator — UHN - Princess Margaret Cancer Centre; Amit Oza, MD, Study Director — Princess Margaret Cancer Centre Drug Development Program
Locations (4):
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

REFERENCES:
- [Background] Bos JL. ras oncogenes in human cancer: a review. Cancer Res. 1989 Sep 1;49(17):4682-9. PMID 2547513
- [Background] Calvert AH. Dose optimisation of carboplatin in adults. Anticancer Res. 1994 Nov-Dec;14(6A):2273-8. PMID 7825958
- [Background] Davies H, Bignell GR, Cox C, Stephens P, Edkins S, Clegg S, Teague J, Woffendin H, Garnett MJ, Bottomley W, Davis N, Dicks E, Ewing R, Floyd Y, Gray K, Hall S, Hawes R, Hughes J, Kosmidou V, Menzies A, Mould C, Parker A, Stevens C, Watt S, Hooper S, Wilson R, Jayatilake H, Gusterson BA, Cooper C, Shipley J, Hargrave D, Pritchard-Jones K, Maitland N, Chenevix-Trench G, Riggins GJ, Bigner DD, Palmieri G, Cossu A, Flanagan A, Nicholson A, Ho JW, Leung SY, Yuen ST, Weber BL, Seigler HF, Darrow TL, Paterson H, Marais R, Marshall CJ, Wooster R, Stratton MR, Futreal PA. Mutations of the BRAF gene in human cancer. Nature. 2002 Jun 27;417(6892):949-54. doi: 10.1038/nature00766. Epub 2002 Jun 9. PMID 12068308
- [Background] Ding L, Getz G, Wheeler DA, Mardis ER, McLellan MD, Cibulskis K, Sougnez C, Greulich H, Muzny DM, Morgan MB, Fulton L, Fulton RS, Zhang Q, Wendl MC, Lawrence MS, Larson DE, Chen K, Dooling DJ, Sabo A, Hawes AC, Shen H, Jhangiani SN, Lewis LR, Hall O, Zhu Y, Mathew T, Ren Y, Yao J, Scherer SE, Clerc K, Metcalf GA, Ng B, Milosavljevic A, Gonzalez-Garay ML, Osborne JR, Meyer R, Shi X, Tang Y, Koboldt DC, Lin L, Abbott R, Miner TL, Pohl C, Fewell G, Haipek C, Schmidt H, Dunford-Shore BH, Kraja A, Crosby SD, Sawyer CS, Vickery T, Sander S, Robinson J, Winckler W, Baldwin J, Chirieac LR, Dutt A, Fennell T, Hanna M, Johnson BE, Onofrio RC, Thomas RK, Tonon G, Weir BA, Zhao X, Ziaugra L, Zody MC, Giordano T, Orringer MB, Roth JA, Spitz MR, Wistuba II, Ozenberger B, Good PJ, Chang AC, Beer DG, Watson MA, Ladanyi M, Broderick S, Yoshizawa A, Travis WD, Pao W, Province MA, Weinstock GM, Varmus HE, Gabriel SB, Lander ES, Gibbs RA, Meyerson M, Wilson RK. Somatic mutations affect key pathways in lung adenocarcinoma. Nature. 2008 Oct 23;455(7216):1069-75. doi: 10.1038/nature07423. PMID 18948947
- [Background] Gervais R, Robinet G, Clement-Duchene C, Denis F, El Kouri C, Martin P, Chouaki N, Bourayou N, Morere JF. Pemetrexed and carboplatin, an active option in first-line treatment of elderly patients with advanced non-small cell lung cancer (NSCLC): a phase II trial. Lung Cancer. 2013 May;80(2):185-90. doi: 10.1016/j.lungcan.2013.01.008. Epub 2013 Feb 21. PMID 23434351
- [Background] Hanna N, Shepherd FA, Fossella FV, Pereira JR, De Marinis F, von Pawel J, Gatzemeier U, Tsao TC, Pless M, Muller T, Lim HL, Desch C, Szondy K, Gervais R, Shaharyar, Manegold C, Paul S, Paoletti P, Einhorn L, Bunn PA Jr. Randomized phase III trial of pemetrexed versus docetaxel in patients with non-small-cell lung cancer previously treated with chemotherapy. J Clin Oncol. 2004 May 1;22(9):1589-97. doi: 10.1200/JCO.2004.08.163. PMID 15117980
- [Background] Janne PA, Shaw AT, Pereira JR, Jeannin G, Vansteenkiste J, Barrios C, Franke FA, Grinsted L, Zazulina V, Smith P, Smith I, Crino L. Selumetinib plus docetaxel for KRAS-mutant advanced non-small-cell lung cancer: a randomised, multicentre, placebo-controlled, phase 2 study. Lancet Oncol. 2013 Jan;14(1):38-47. doi: 10.1016/S1470-2045(12)70489-8. Epub 2012 Nov 28. PMID 23200175
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Juergens RA, Brahmer JR. Adjuvant treatment in non-small cell lung cancer: Where are we now? J Natl Compr Canc Netw. 2006 Jul;4(6):595-600. doi: 10.6004/jnccn.2006.0049. PMID 16813727
- [Background] Kwak EL, Bang YJ, Camidge DR, Shaw AT, Solomon B, Maki RG, Ou SH, Dezube BJ, Janne PA, Costa DB, Varella-Garcia M, Kim WH, Lynch TJ, Fidias P, Stubbs H, Engelman JA, Sequist LV, Tan W, Gandhi L, Mino-Kenudson M, Wei GC, Shreeve SM, Ratain MJ, Settleman J, Christensen JG, Haber DA, Wilner K, Salgia R, Shapiro GI, Clark JW, Iafrate AJ. Anaplastic lymphoma kinase inhibition in non-small-cell lung cancer. N Engl J Med. 2010 Oct 28;363(18):1693-703. doi: 10.1056/NEJMoa1006448. PMID 20979469
- [Background] Maione P, Gridelli C, Troiani T, Ciardiello F. Combining targeted therapies and drugs with multiple targets in the treatment of NSCLC. Oncologist. 2006 Mar;11(3):274-84. doi: 10.1634/theoncologist.11-3-274. PMID 16549812
- [Background] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680
- [Background] Okamoto I, Aoe K, Kato T, Hosomi Y, Yokoyama A, Imamura F, Kiura K, Hirashima T, Nishio M, Nogami N, Okamoto H, Saka H, Yamamoto N, Yoshizuka N, Sekiguchi R, Kiyosawa K, Nakagawa K, Tamura T. Pemetrexed and carboplatin followed by pemetrexed maintenance therapy in chemo-naive patients with advanced nonsquamous non-small-cell lung cancer. Invest New Drugs. 2013 Oct;31(5):1275-82. doi: 10.1007/s10637-013-9941-z. Epub 2013 Mar 10. PMID 23475281
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Pao W, Girard N. New driver mutations in non-small-cell lung cancer. Lancet Oncol. 2011 Feb;12(2):175-80. doi: 10.1016/S1470-2045(10)70087-5. PMID 21277552
- [Background] Scagliotti GV, Parikh P, von Pawel J, Biesma B, Vansteenkiste J, Manegold C, Serwatowski P, Gatzemeier U, Digumarti R, Zukin M, Lee JS, Mellemgaard A, Park K, Patil S, Rolski J, Goksel T, de Marinis F, Simms L, Sugarman KP, Gandara D. Phase III study comparing cisplatin plus gemcitabine with cisplatin plus pemetrexed in chemotherapy-naive patients with advanced-stage non-small-cell lung cancer. J Clin Oncol. 2008 Jul 20;26(21):3543-51. doi: 10.1200/JCO.2007.15.0375. Epub 2008 May 27. PMID 18506025
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Schuette WH, Groschel A, Sebastian M, Andreas S, Muller T, Schneller F, Guetz S, Eschbach C, Bohnet S, Leschinger MI, Reck M. A randomized phase II study of pemetrexed in combination with cisplatin or carboplatin as first-line therapy for patients with locally advanced or metastatic non-small-cell lung cancer. Clin Lung Cancer. 2013 May;14(3):215-23. doi: 10.1016/j.cllc.2012.10.001. Epub 2013 Jan 16. PMID 23332288
- [Background] Spira A, Ettinger DS. Multidisciplinary management of lung cancer. N Engl J Med. 2004 Jan 22;350(4):379-92. doi: 10.1056/NEJMra035536. No abstract available. PMID 14736930
- [Background] Zukin M, Barrios CH, Pereira JR, Ribeiro Rde A, Beato CA, do Nascimento YN, Murad A, Franke FA, Precivale M, Araujo LH, Baldotto CS, Vieira FM, Small IA, Ferreira CG, Lilenbaum RC. Randomized phase III trial of single-agent pemetrexed versus carboplatin and pemetrexed in patients with advanced non-small-cell lung cancer and Eastern Cooperative Oncology Group performance status of 2. J Clin Oncol. 2013 Aug 10;31(23):2849-53. doi: 10.1200/JCO.2012.48.1911. Epub 2013 Jun 17. PMID 23775961
- [Derived] Fung AS, Graham DM, Chen EX, Stockley TL, Zhang T, Le LW, Albaba H, Pisters KM, Bradbury PA, Trinkaus M, Chan M, Arif S, Zurawska U, Rothenstein J, Zawisza D, Effendi S, Gill S, Sawczak M, Law JH, Leighl NB. A phase I study of binimetinib (MEK 162), a MEK inhibitor, plus carboplatin and pemetrexed chemotherapy in non-squamous non-small cell lung cancer. Lung Cancer. 2021 Jul;157:21-29. doi: 10.1016/j.lungcan.2021.05.021. Epub 2021 May 24. PMID 34052705
- See also: Publication — https://doi.org/10.1016/j.lungcan.2021.05.021

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled based on physician referral, 1st participant was enrolled on 07 March 2017 and last participant was enrolled on 05 December 2018
Pre-assignment Details: Out of 16 patients screened, 13 were enrolled who met the eligibility criteria
Groups:
- Binimetinib Dose Level 1 (30mg BID): Phase I, dose level 1 group:
  The dose of MEK162 for dose level 1 group will be 30 mg BID.
  Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Minimum number of patients is 3.
  The rate of subject entry and escalation to the next dose level will depend upon assessment of the safety profile of patients entered at the previous dose level.
- Binimetinib Dose Level 2 (45mg BID): Phase I, dose level 2 group:
  The dose of MEK162 for dose level 2 group will be 45 mg BID. Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Minimum number of patients is 3. The rate of subject entry and escalation to the next dose level will depend upon assessment of the safety profile of patients entered at the previous dose level.
Period: Binimetinib Dose Level 1 (30mg BID)
Arm/Group | Binimetinib Dose Level 1 (30mg BID) | Binimetinib Dose Level 2 (45mg BID)
Started | 6 | 0 (One patient was not evaluable for DLT; therefore, an additional patient was enrolled at DL2)
Completed | 6 | 0 (One patient was not evaluable for DLT; therefore, an additional patient was enrolled at DL2)
Not Completed | 0 | 0
Period: Binimetinib Dose Level 2 (45mg BID)
Arm/Group | Binimetinib Dose Level 1 (30mg BID) | Binimetinib Dose Level 2 (45mg BID)
Started | 0 | 7
Completed | 0 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients 18 years or older with histologically confirmed stage IV non squamous NSCLC were eligible. Patients were treated with binimetinib in combination with first-line carboplatin and pemetrexed chemotherapy.
Groups:
- Binimetinib Dose Level 1: Phase I, dose level 1 group:
  The dose of MEK162 for dose level 1 group will be 30 mg BID.
  Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Minimum number of patients is 3.
  The rate of subject entry and escalation to the next dose level will depend upon assessment of the safety profile of patients entered at the previous dose level.
- Binimetinib Dose Level 2: Phase I, dose level 2 group:
  The dose of MEK162 for dose level 2 group will be 45 mg BID. Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Minimum number of patients is 3. The rate of subject entry and escalation to the next dose level will depend upon assessment of the safety profile of patients entered at the previous dose level.
- Binimetinib Dose Level -1: Dose de-escalation group:
  The dose of MEK162 for dose level -1 group will be 30 mg BID. Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Minimum number of patients is 3. The rate of subject entry and escalation or de-escalation will depend upon assessment of the safety profile of patients and dose limiting toxicities.
- Total: Total of all reporting groups
Arm/Group | Binimetinib Dose Level 1 | Binimetinib Dose Level 2 | Binimetinib Dose Level -1 | Total
Number analyzed (Participants) | 6 | 7 | 0 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 0 | 9
  >=65 years | 2 | 2 | 0 | 4
Age, Continuous [Median (Full Range); unit: years] | 63.166 [50 to 81] | 56.428 [42 to 74] |  | 59.538 [42 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 |  | 6
  Male | 2 | 5 |  | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 7 |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose in Milligrams Per Day for Binimetinib.
Description: To determine the recommended dose in milligrams per day of the combination of MEK162 with standard therapy pemetrexed and carboplatin as determined by toxicity.
Time Frame: 22 weeks
Population: One patient was not evaluable for DLT; therefore, an additional patient was enrolled at Dose Level 2.
  The outcome measure for the recommended does is 30 mg, both arms were combined in the analysis here in order to report 1 recommended single dose (30mg).
Measure: Number; unit: mg
Groups:
- Binimetinib Dose Level 1 & 2 (30mg BID & 45mg BID): Phase I, dose level 1 & 2 groups:
  The dose of MEK162 for dose level 1 group will be 30 mg BID and for dose level 2 will be 45 mg BID.
  Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
Arm/Group | Binimetinib Dose Level 1 & 2 (30mg BID & 45mg BID)
Number analyzed (Participants) | 12
mg | 30

2. Secondary Outcome: Objective Response Rate (ORR) as Per RECIST v1.1.
Description: The size of tumors in centimeters before and after treatment. The measurements will be compared against the RECIST v1.1 criteria to ascertain response as defined in the protocol.
  Objective response rate (ORR) was defined as the percentage of patients who achieved a complete or partial response as the best overall response.
Time Frame: 22 weeks
Population: Objective response rate (ORR) was defined as the percentage of patients who achieved a complete or partial response as the best overall response.
Measure: Count of Participants; unit: Participants
Groups:
- Binimetinib Dose Level 1 (30mg BID): 4/6 patients achieved partial response for Dose Level 1 (67%)
- Binimetinib Dose Level 2 (45mg BID): Dose level 2 arm had 7 patients but 1 was non-evaluable, so 6 patients only were evaluable.
  2/6 patients achieved partial response for Dose Level 2 (33%)
Arm/Group | Binimetinib Dose Level 1 (30mg BID) | Binimetinib Dose Level 2 (45mg BID)
Number analyzed (Participants) | 6 | 6
Participants | 4 | 2

3. Other Pre Specified Outcome: Exploratory Analysis of Objective Response Rate, KRAS Mutation Sub-type.
Description: Exploratory analysis of mutation subtypes using next generation sequencing (NGS).
Time Frame: 22 weeks
Population: Dose levels are combined as mutation information was obtained for the 12 patients in total and segregated in the results by these 2 groups only. Link to published results/ https://doi.org/10.1016/j.lungcan.2021.05.021
Measure: Number; unit: percentage of participants
Groups:
- KRAS/NRAS-mutated Patients: Exploratory analysis of KRAS/NRAS-mutated patients.
- KRAS/NRAS Wild-type Patients: Exploratory analysis of KRAS/NRAS wild-type patients.
Arm/Group | KRAS/NRAS-mutated Patients | KRAS/NRAS Wild-type Patients
Number analyzed (Participants) | 7 | 5
percentage of participants | 62.5 | 25

4. Other Pre Specified Outcome: Progression Free Survival Rate
Description: Evaluation progression-free survival rate (PFS) for patients with and without KRAS mutation in tumor tissue. PFS is defined as the time from start of treatment to disease progression or death.
  PFS rate is measured over 6 months period (26 weeks). PFS rate is calculated as a percentage of participants achieving a 6 months (26 weeks) period of progression free survival.
Time Frame: 26 weeks
Population: Phase Ib. Evaluation of progression-free survival (PFS) rate for patients with and without KRAS mutation in tumor tissue. PFS is defined as the time from start of treatment to disease progression or death.
  PFS rate is calculated as a percentage of participants achieving a 6 months (26 weeks) period of progression free survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall Study Progression Free Survival Rate: Progression free survival (PFS) was defined as the time from the start of treatment to the time of progression or death.
Arm/Group | Overall Study Progression Free Survival Rate
Number analyzed (Participants) | 12
percentage of participants | 38.5 [19.3 to 76.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were recorded for 22 weeks of treatment.
Description: An adverse event is any untoward medical occurrence (including any abnormal laboratory finding), symptom, or disease temporarily associated with the use of a medicinal (investigational product) in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with treatment.
  Plus Expected Adverse Events and SAEs for MEK162 as per protocol. Systematic Assessment: Through standard questionnaire, regular PI assessment and regular lab testing.
Groups:
- Binimetinib Dose Level -1 (30mg BID): Dose de-escalation group:
  The dose of MEK162 for dose level -1 group will be 30 mg BID. Carboplatin will be given every 3 weeks. Pemetrexed will be given every 3 weeks.
  Pemetrexed: 4-6 cycles given intravenously in combination with carboplatin as per standard therapy.
  Carboplatin: 4-6 cycles of intravenous Carboplatin in combination with Pemetrexed as per standard therapy.
  Minimum number of patients is 3. The rate of subject entry and escalation or de-escalation will depend upon assessment of the safety profile of patients and dose limiting toxicities.
Arm/Group | Binimetinib Dose Level 1 (30mg BID) | Binimetinib Dose Level 2 (45mg BID) | Binimetinib Dose Level -1 (30mg BID)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/7 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 3/7 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Binimetinib Dose Level 1 (30mg BID) (N=6) | Binimetinib Dose Level 2 (45mg BID) (N=7) | Binimetinib Dose Level -1 (30mg BID) (N=0)
Diverticulitis (grade 3) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (grade 3) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary infection (grade 2) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (grade 3) (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — patient admitted with confusion felt to be unrelated to treatment.
Cerebral metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) — patient died from progression of cerebral metastases.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Binimetinib Dose Level 1 (30mg BID) (N=6) | Binimetinib Dose Level 2 (45mg BID) (N=7) | Binimetinib Dose Level -1 (30mg BID) (N=0)
ALT Increase (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
AST Increase (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bilateral Leg Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bilirubin Increase (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Dry skin/Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 0 (0)
Dysuria/Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 3 (3) | 2 (2) | 0 (0)
Ejection Fraction Decrease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Mucositis (Oral, Nasal) (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
Neutrophil Count Decrease (Immune system disorders) | 2 (2) | 2 (2) | 0 (0)
Ocular toxicity (Eye disorders) | 5 (5) | 3 (3) | 0 (0)
Palpitations/Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Serum Amylase Increase (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Weight Gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Decrease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT02185690/Prot_SAP_000.pdf